CLINICAL TRIAL: NCT01846312
Title: The Longitudinal Diabetes Biomarker Study: An Observational Study to Assess Longitudinal Variation of Immune Biomarkers in Subjects at Risk for Development of Type 1 Diabetes
Brief Title: An Observational Study to Assess Longitudinal Variation of Immune Biomarkers in Subjects at Risk for Development of Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4074; U1111-1136-8383 (Other: WHO)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling for biomarkers. A portion of each sample collected will be tested for five different islet autoantibodies (presence and precise titers). The remaining portion of each sample will be coded and then assessed for autoantibody isotypes, phenotyping of peripheral blood mononuclear cells (PBMC), and profiling of cytokines, and pharmacogenetic markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The participants will not receive any treatment.

SUMMARY:
This study is conducted in the United States of America (USA). The aim of the study is to assess longitudinal variation of immune biomarkers in subjects at risk for development of type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with general good health as judged by the investigator
* Participant tested positive at above or equal to 99th percentile for one or more of three islet antibodies (GAD (glutamic acid decarboxylase), IA2 (islet antigen-2), IAA (insulin autoantibody))

Exclusion Criteria:

* Any chronic disorder (diabetes at enrolment) or severe disease which, in the opinion of the investigator, might jeopardize subject's safety or compliance with the protocol
* Female of child-bearing potential who is pregnant, breast-feeding, or intends to become pregnant

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects who are at risk for developing T1D either by genetic testing or due to family history and identified with one or more islet autoantibodies).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fluctuation in islet autoantibodies titers | One-two years dependent on sampling frequency

SECONDARY OUTCOMES:
Fluctuation in islet autoantibody isotypes | One-two years dependent on sampling frequency
Fluctuation in T-cell specificity profiling (mainly for CD8 (cluster of differentiation 8) T-cells) | One-two years dependent on sampling frequency

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com